CLINICAL TRIAL: NCT04613661
Title: Inter-rater Reliability of the Australian Spasticity Assessment Scale (ASAS) in Post-stroke Spasticity
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ilker şengül, Principal Investigator, Izmir Katip Celebi University
Other Study IDs: 2020-GOKAE-0450
Record Dates: First submitted 2020-10-23; First posted 2020-11-03 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Hemiplegia, Spastic
Keywords: Hemiplegia; spasticity; upper limb
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Researcher 1: The first researcher assessing elbow, wrist, and ankle spasticity, respectively
  Interventions: Other: Australian Spasticity Assessment Scale
- Researcher 2: The second researcher assessing elbow, wrist, and ankle spasticity, respectively
  Interventions: Other: Australian Spasticity Assessment Scale

INTERVENTIONS:
Other: Australian Spasticity Assessment Scale — Australian Spasticity Assessment Scale is a clinical measure to assess the severity of spasticity

SUMMARY:
The reliability of the Australian Spasticity Assessment Scale (ASAS) has been reported to be not high enough in adult patients with acquired brain damage. The low number of patients and the heterogeneous study population have been reported as important limitations in the reliability study of this measure. Therefore, the reliability of the ASAS needs to be confirmed in stroke patients with spasticity. This study aims to investigate the inter-rater reliability of the ASAS in a study population consisting of a larger and more homogeneous patient population (those with post-stroke spasticity).

DETAILED DESCRIPTION:
Spasticity is a motor disorder characterized by a velocity-dependent increase in tonic stretch reflex due to upper motor neuron lesion. The prevalence of post-stroke spasticity is between 17-40%. In the assessment of spasticity, although biomechanical and neurophysiological methods provide quantitative data, semi-quantitative methods are mostly used clinically. The most frequently used spasticity measures are the Modified Ashworth Scale and the Modified Tardieu Scale. However, these methods have significant disadvantages. Therefore, the search for more reliable clinical measures continues. One of the newly developed clinical scales is called the Australian Spasticity Assessment Scale (ASAS). Although ASAS has been reported to have a high level of reliability in children with cerebral palsy, the same has not been detected in adult patients with acquired brain damage. The low number of patients and the heterogeneous study population have been reported as two of the important limitations in the reliability study of this measure.

In this study, researchers aim to investigate the inter-rater reliability of the ASAS in a study population consisting of a larger and more homogeneous patient population (those with post-stroke spasticity).

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke (> 6 months)
* Fist stroke
* Increased tone according to the Modified Ashworth Scale in at least one of the elbow, wrist, and ankle
* Stability of spasticity for the last 3 months

Exclusion Criteria:

* Increased tone due to causes other than stroke (traumatic brain injury, spinal cord injury, multiple sclerosis, motor neuron disease, etc.)
* Acute or subacute stroke (≤6 months)
* Recurrent stroke attacks
* Presence of contracture and/or moderate to severe pain in the joints to be assessed (elbow, wrist, and ankle)
* Botulinum toxin injection in the last three months
* History of neurolysis for spasticity (alcohol or phenol)
* History of surgery for spasticity
* Initiation of a new drug for spasticity, or a change in drug dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic stroke patients with elbow and/or wrist and /or ankle spasticity
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Australian Spasticity Assessment Scale (ASAS) | Through study completion, an average of 2 year
  The ASAS is an ordinal scale with five levels (0, 1, 2, 3, 4). The severity of spasticity increases as the level-ups.The contracture is assessed separately. Level 0 means no catch on rapid passive stretch (no spasticity), and level 4 means that the body part is fixed on the rapid passive stretch but moves on the slow passive stretch. In level 1, a catch followed by a release occurs on the rapid passive stretch. In level 2, the catch is in the second half of the range, and there is a resistance in the remaining range of motion. In level 3, the catch is in the first half of the range, and there is a resistance in the remaining range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: İlker Şengül, M.D., Principal Investigator — İzmir Katip Çelebi University
Locations (1):
- İlker Şengül, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lance JW. The control of muscle tone, reflexes, and movement: Robert Wartenberg Lecture. Neurology. 1980 Dec;30(12):1303-13. doi: 10.1212/wnl.30.12.1303. No abstract available. PMID 7192811
- [Background] Lundstrom E, Terent A, Borg J. Prevalence of disabling spasticity 1 year after first-ever stroke. Eur J Neurol. 2008 Jun;15(6):533-9. doi: 10.1111/j.1468-1331.2008.02114.x. Epub 2008 Mar 18. PMID 18355307
- [Background] Wissel J, Manack A, Brainin M. Toward an epidemiology of poststroke spasticity. Neurology. 2013 Jan 15;80(3 Suppl 2):S13-9. doi: 10.1212/WNL.0b013e3182762448. PMID 23319481
- [Background] Pierson SH. Outcome measures in spasticity management. Muscle Nerve Suppl. 1997;6:S36-60. PMID 9826982
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Love S, Gibson N, Smith N, Bear N, Blair E; Australian Cerebral Palsy Register Group. Interobserver reliability of the Australian Spasticity Assessment Scale (ASAS). Dev Med Child Neurol. 2016 Feb;58 Suppl 2:18-24. doi: 10.1111/dmcn.13000. Epub 2016 Jan 14. PMID 26762706
- [Background] Calame A, Singer B. Inter- and Intra-Rater Reliability of the Australian Spasticity Assessment Scale in Adults with Acquired Brain Injury. Open Journal of Therapy and Rehabilitation. 2015;3:77-86.